CLINICAL TRIAL: NCT04416113
Title: Photobiomodulation and Photodynamic Therapy for the Treatment of COVID-19 A Randomized Controlled Clinical Trials
Brief Title: Photodynamic Therapy for the Treatment of COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abeer Attia Tawfik, professor of dermatology and laser at national institute of laser enhanced sciences, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cu-NILES/16/20
Record Dates: First submitted 2020-05-24; First posted 2020-06-04 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Photodynamic Therapy& Low Level Laser in Management of COVID 19
Keywords: photodynamic therapy; low level laser therapy; COVID 19 virus
MeSH Terms: interventions — Low-Level Light Therapy; Photochemotherapy; Congresses as Topic

STUDY DESIGN:
Intervention Model Description: A randomized controlled study will be conducted on 60 patients of positive COVID 19. The patients will be divided into 3 equal groups. Group I will receive low level laser (diode laser 980nm) from laser watch for 30 minutes, 20 J for 3 to 5 days and laser acupuncture. Group 2 will be treated with photodynamic therapy by injecting the methylene blue as a photosensitizer and irradiated with laser watch (diode laser 670 nm). Group 3 will serve as a control. Evaluation methods will include laboratory investigations and CT chest.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- photobiomodulation group (Active Comparator): Laser watch Patients will be subjected to low-level laser (diode laser 980nm) for 30 minutes, the recommended dose based on the previous study is 20 J for 3 to 7 days.
  The laser device:
  Laser watched applied at the wrist on the radial artery.
  Laser acupuncture
  Interventions: Procedure: photobiomodulation and photodynamic therapy
- photodynamic group (Active Comparator): Methylene blue injection USP 1% will be used as a photosensitizer in PDT.
  * 0.1 to 0.2 mL of 1% solution per kilogram of body weight Methylene Blue (methylene blue injection) will be injected intravenously very slowly over a period of several minutes to
  * After one hour apply Light dose: 100 - 200 J/cm2 50-100 mW/cm2. (50 mW/cm2 increased the phototoxic response as well as the fractionated light application).
  * The session will be done twice per week
  Laser watched applied at the wrist on the radial artery.
  Interventions: Procedure: photobiomodulation and photodynamic therapy
- positive control (Active Comparator): This group will include patients who are subjected to conventional treatment
  Interventions: Procedure: photobiomodulation and photodynamic therapy

INTERVENTIONS:
Procedure: photobiomodulation and photodynamic therapy — antiviral treatment
  Other Names: conventional

SUMMARY:
Until now there is no vaccine or reliable treatment for the COVID-19 pandemic. The fundamental mechanisms of non-invasive low-level laser in photobiomodulation (PBM) and photodynamic therapy is to stimulate the mitochondrial respiratory chain where a transient release of non-cytotoxic levels of reactive oxygen species (ROS) will lead to positive modulation of the immune response. As previous studies mentioned that the most important strategy for COVID-19 management is oxygenation and faster rehabilitation of the damaged tissue, antiviral effects, and, ﬁnally, reduction or controlling the cytokine storm by reducing inﬂammatory agents. PBM may be used as adjuvant therapy or even an alternative therapy in all these mechanisms without side effects and drug interactions.

Objectives The objective of this clinical trial is to use the photobiomodulation therapy (PBMT), and photodynamic therapy as adjuvant therapy or even an alternative therapy for Covide-19.

Patients and methods A randomized controlled study will be conducted on 60 patients of positive COVID 19. The patients will be divided into 3 equal groups. Group, I will receive a low-level laser (diode laser 980nm) from laser watch for 30 minutes, 20 J for 3 to 5 days, and laser acupuncture. Group 2 will be treated with photodynamic therapy by injecting the methylene blue as a photosensitizer and irradiated with laser watch (diode laser 670 nm). Group 3 will serve as a control. Evaluation methods will include laboratory investigations and CT chest.

DETAILED DESCRIPTION:
Treatment protocol:

This clinical study was conducted following the approval of the research ethics committee for experimental and clinical studies at the National Institute of Laser Enhanced Sciences, Cairo University, Egypt (approval number CU-NILES/16/20 May 2020) with the principles outlined in the Declaration of Helsinki for human subject experimentation being followed. Informed consent will be obtained from the patients, and the privacy rights will be continuously observed.

This study will be conducted on 60 patients with COVID 19 of all ages and both sex.

Patients will be divided into 3 groups:

Group 1: photobiomodulation This group included the use of laser watch and laser acupuncture

Laser watch Patients will be subjected to low level laser (diode laser 980nm) for 30 minutes, the recommended dose based on previous study is 20 J for 3 to 7 days.

The laser device:

Laser watched applied at the wrist on the radial artery.

Laser acupuncture Patients will receive laser acupuncture using pulsed infra- red laser, wavelength 880 / 905/980 nm, spot size diameter of 5 mm frequency 2500 Hz, average power 15 W, energy of 225 mJ applied for 2 min per point and pulse width of 100 ns and area = 0.2 cm2. Patients will receive one session daily for 7 days.

Laser acupuncture was applied at the following points (World Health Organization 2008). The points where the laser acupuncture will be applied are demonstrated in the following figures:

* For cough and chest tightness, wheezes and congestion: LU1, 2, 5, 7, 9, 14 (fig.1) For improving immunity and blood circulation, also for dyspnea and GIT manifestation also, breaks up blood stagnation in the chest: ST36
* Affects the throat, chest, lungs: CV12, CV4 Sore throat, coughing, & asthma: KI3 Fig
* Laser acupuncture device could be applied simultaneously on all points same time by special multi-channel device (fig3)

Group 2 (photodynamic therapy) Methylene blue injection USP 1% will be used as a photosensitizer in PDT.

* 0.1 to 0.2 mL of 1% solution per kilogram of body weight Methylene Blue (methylene blue injection) will be injected intravenously very slowly over a period of several minutes to prevent local high concentration of the compound from producing methemoglobin (low concentrations will convert methemoglobin to hemoglobin and will be activated by light).
* After one hour apply Light dose: 100 - 200 J/cm2 50-100 mW/cm2. (50 mW/cm2 increased the phototoxic response as well as fractionated light application).
* Session will be done twice per week

The laser device:

Laser watched applied at the wrist on the radial artery. Group 3: positive control This group will include patients who are subjected to conventional treatment Evaluation and assessment All patients will be subjected to thorough examination with complete personal and clinical history and will do the following before and after treatment: PCR, CBC, CRP, ESR, D dimers, liver enzymes, and Ferritin, CT chest

Endpoint Treatment will be stopped if no improvement occurred after one week

Statistical analysis

All statistical calculations were done using computer programs SPSS (Statistical Package for the Social Science; SPSS Inc., Chicago, IL) v.16 for Microsoft Windows. Continuous variables were tested for normality by the Shapiro-Wilk normality test. Values are presented as mean ± standard deviation, or in the case of non-normally distributed data as median and inter-quartile range. For comparison between paired parameters (before and after treatment), paired t-test or the Wilcoxon matched-pairs signed-rank test were used according to data normality. For comparison between independent groups, the chi-squared test was used to compare percentages between different groups of patients. Normally distributed data were analyzed using independent samples t-test. Non-normally distributed data were analyzed using the Mann-Whitney U-test. p values <.05 were considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with Positive COVID 19 test suffering from Fever, cough, shortness of breath, chills, muscle pain, the new loss of taste or smell, vomiting or diarrhea, and/or sore throat

Exclusion Criteria:

* Patients in critical cases who admitted to the ICU, bacterial pneumonia, and respiratory distress grade III, IV, and patients on a mechanical ventilator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-08-05 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Participants Achieving Either a Major Clinical Response or Partial Clinical Response (PCR) Defined by WHO | 2 weeks
  Molecular-based assays:
  * N COV 2019
  * Antigen assays:
  * SARS (COV) antigen, Serology assays:
  * N COV 2019 antibodies medical respiratory clearance questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Abeer Attia Tawfik, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No
if the results are positive we will invite other researchers to share

REFERENCES:
- [Background] Mahase E. Covid-19: what treatments are being investigated? BMJ. 2020 Mar 26;368:m1252. doi: 10.1136/bmj.m1252. No abstract available. PMID 32217607
- [Background] Fekrazad R. Photobiomodulation and Antiviral Photodynamic Therapy as a Possible Novel Approach in COVID-19 Management. Photobiomodul Photomed Laser Surg. 2020 May;38(5):255-257. doi: 10.1089/photob.2020.4868. Epub 2020 Apr 23. No abstract available. PMID 32326830